CLINICAL TRIAL: NCT01407718
Title: The Parapatellar Approach to Intramedullary Tibial Nailing: Is There a Difference in Anterior Knee Pain When Compared to a Traditional Flexed Approach?
Brief Title: The Parapatellar Approach to Intramedullary Tibial Nailing
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Rothberg, M.D., University of Utah
Other Study IDs: 43060
Record Dates: First submitted 2011-07-27; First posted 2011-08-02 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Knee Pain Intermittent
Keywords: Knee pain; tibial nailing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will address the incidence of anterior knee pain in the approaches used for tibial nailing. A parapatellar approach, with nail insertion in relative extension, will be compared to the approaches in which nail insertion requires the knee to be placed in flexion. The incidence of anterior knee pain will be compared in each group to assess whether the compared approaches result in similar levels of anterior knee pain. Patients will be given the 2000 IKDC Subjective Knee Evaluation Form to assess anterior knee pain. The 2000 IKDC Subjective Knee Evaluation Form is a newer assessment tool created by the International Knee Documentation Committee. It has been validated for use with broad patient populations dealing with various knee disorders.19

DETAILED DESCRIPTION:
In the population affected by orthopaedic injury, fractures of the tibial shaft are the most common of all long bone fractures. This fracture pattern occurs approximately 26 times per 100,000 people and accounts for 77,000 hospitalizations per annum.(1, 2) Intramedullary nailing is the most common operative treatment choice for fractures of the diaphyseal tibia (tibial shaft). Intramedullary nailing is also commonly used for shaft fractures that extend into the metaphyses (excluding fractures that extend into the knee and/or exhibit comminution at the ankle joint).

Tibial nails are inserted at or about the knee. Three different insertion approaches are used as standard of care at this institution, including the transtendinous, peritendinous, and parapatellar approach. In all three techniques, the nail is placed in the tibia in the same manner: after fracture reduction, the proper entry point in the proximal tibia is found and the tibia is sequentially reamed until a suitable nail can be passed and locked in place with interlocking screws. The three named approaches vary the (1) angulation of the knee at the time of insertion and the (2) location of the incision and soft tissue dissection, relative to the patellar tendon, necessary to locate the proper entry point for the nail. Tibial nails are inserted with the knee in flexion (bent to ~90°) for the transtendinous and peritendinous approaches, and in relative extension (less than 30°) for the parapatellar approach. For insertion, the transtendinous and peritendinous approaches require dissections that allow the nail to be passed through or around the patellar tendon. In the parapatellar technique, dissection is carried out juxtaposed to the patella.

Anterior knee pain is the most common complication of intramedullary tibial nailing. It has been reported in a range of 10% to 86% with average follow up of two years.(3) Review of current literature regarding the subject of anterior knee pain and tibial nailing reveals four commonly attributable causes: skin incision location,(4,5) approach in reference to the patellar tendon,(6-9) nail insertion site,(10) and nail prominence.(11-13) No study has specifically examined whether knee angulation at the time of insertion impacts anterior knee pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years of age or older, who present to the University of Utah Medical Center for treatment of a tibia fracture that requires use of an intramedullary nail for fracture fixation.

Exclusion Criteria:

* prior operations about the knee
* neurovascular compromise
* ipsilateral fracture of the femur or proximal tibia not amenable to intramedullary nailing
* patients who are non-ambulatory
* patients who have ipsilateral fractures involving the ankle or foot
* a fracture pattern that requires the surgeon to use a surgical approach outside the assigned treatment arm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be indicated for intramedullary tibial nailing according to their fracture pattern.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
incidence of anterior knee pain in the approaches used for tibial nailing | 6 months after surgery
  This project will address the incidence of anterior knee pain in the approaches used for tibial nailing. A parapatellar approach, with nail insertion in relative extension, will be compared to the approaches in which nail insertion requires the knee to be placed in flexion

SECONDARY OUTCOMES:
compare knee pain levels in patients whose tibial fractures required intramedullary nailing and were treated using a parapatellar approach | 1 year after surgery
  The purpose of this prospective study is to compare knee pain levels in patients whose tibial fractures required intramedullary nailing and were treated using a parapatellar approach (knee flexed ~30 degrees) or a traditional approach requiring full flexion of the knee (transtendinous and peritendinous approaches utilize flexion of ~90 degrees).

CONTACTS AND LOCATIONS:
Overall Officials: David Rothberg, MD, Principal Investigator — University of Utah Orthapedics
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States